CLINICAL TRIAL: NCT05529108
Title: Impact of Brewer's Spent Grain (BSG) and Bio-transformed BSG Biscuits on Glycaemic Control and Gut Health in Singapore Adults With Metabolic Syndrome
Brief Title: Glycaemic Control Effect of BSG and Underlying Gut - Related Mechanism in Singapore Adults With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S20
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome; Diabetes
Keywords: Metabolic Syndrome; middle-aged and older adults; Post-prandial Glycaemic response; bio-transformed food
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control biscuits group (Placebo Comparator): Subjects are required to consume 90 g control biscuits as their breakfast everyday during 12-week intervention period.
  Interventions: Dietary Supplement: control biscuits
- autoclaved BSG-containing group (Experimental): Subjects are required to consume 90 g autoclaved BSG-containing biscuits as their breakfast everyday during 12-week intervention period.
  Interventions: Dietary Supplement: autoclaved BSG-containing biscuits
- bio-transformed BSG-containing group (Experimental): Subjects are required to consume 90 g fermented BSG-containing biscuits as their breakfast everyday during 12-week intervention period.
  Interventions: Dietary Supplement: bio-transformed BSG-containing biscuits

INTERVENTIONS:
Dietary Supplement: control biscuits — Consumption of plain biscuits everyday during intervention period.
  Arms: Control biscuits group
Dietary Supplement: autoclaved BSG-containing biscuits — Consumption of autoclaved BSG-containing biscuits everyday during intervention period.
  Arms: autoclaved BSG-containing group
Dietary Supplement: bio-transformed BSG-containing biscuits — Consumption of bio-transformed BSG-containing biscuits everyday during intervention period.
  Arms: bio-transformed BSG-containing group

SUMMARY:
The purpose of this research project is to assess the glycaemic controlling effects of consuming BSG and bio-transformed BSG-containing biscuits and its underlying gut - related mechanism in adults with MetS using in-vivo setting.

DETAILED DESCRIPTION:
This is a double-blind, randomised, parallel experiment, all subjects (38 adults in Singapore with MetS) will complete a 12-week intervention period. Subjects will be randomly assigned to consume their habitual diet with biscuit that either does not contain or contains autoclaved BSG or bio-transformed BSG for 12 weeks. Throughout the intervention, subjects will be assessed for glucose, insulin, lipid and amino acid responses, biomarkers of gut health, and as well as other markers of health.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, aged 35-85 years old
* English-literate and able to give informed consent in English
* Willing to follow the study procedures
* Meet any 3 of the 5 following NCEP-ATP III MetS criteria: waist circumference > 102 cm (male), > 88 cm (female) (For Asian population: Waist circumference > 90 cm (male), > 80 cm (female)); fasting glucose concentration ≥ 100 mg/dL or on medication; triglyceride ≥ 150 mg/dL or on medication; high density lipoprotein cholesterol (HDL) < 40 mg/dL (male), < 50 mg/dL (female); systolic or diastolic blood pressure > 130/85 mmHg or on medication);

Exclusion Criteria:

* Significant change in weight (≥ 3 kg body weight) during the past 3 months
* Allergy to barley, wheat, corn, egg, or other ingredients found inside the biscuits.
* Acute illness at the study baseline
* Exercising vigorously* over the past 3 months. *Defined as having > 6 metabolic equivalents of exercise daily; approximately 20 mins of moderate intensity exercise (e.g. slow jogging) a day
* Following any restricted diet (e.g. vegetarian)
* Smoking
* Have a daily intake of more than 2 alcoholic drinks per day
* Taking dietary supplements or food which may impact the outcome of interests (e.g. fermented foods, probiotic supplement etc.)
* Consumption of antibiotics over past 3 months.
* Pregnant, lactating, or planning pregnancy in the next 6 months
* Insufficient venous access to allow the blood collection
* Prescribed and taking antihypertensive/cholesterol-lowering/ type-2 diabetic medication which started less than 3 years prior to the intervention participation
* High current intake of fibre* from brown rice or wholemeal products. *High, moderate or low intake taken as ≥ 6 servings, 4 - 5 servings, and ≤ 3 servings daily respectively based on My Healthy Plate guidelines
* High current intake of fibre* from vegetables. * High, moderate or low intake taken as ≥ 2 servings, 2 servings, and ≤ 1 serving respectively based on My Healthy Plate guidelines

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose concentration | Every 12 week (week 0 and week 12)
  Glucose concentration in the blood will be measured
Change in insulin concentration | Every 12 week (week 0 and week 12)
  Insulin concentration in the blood will be measured
Change in blood triglyceride concentration | Every 12 week (week 0 and week 12)
  Triglyceride concentration in the blood will be measured
Change in blood cholesterol concentration | Every 12 week (week 0 and week 12)
  Total cholesterol concentration in the blood will be measured
Change in blood Low-density Lipoprotein-cholesterol (LDL) concentration | Every 12 week (week 0 and week 12)
  Low-density Lipoprotein-cholesterol concentration in the blood will be measured
Change in High-density Lipoprotein-cholesterol (HDL) concentration | Every 12 week (week 0 and week 12)
  High-density Lipoprotein-cholesterol concentration in the blood will be measured
Change in Hemoglobin A1c (HbA1c) concentration | Every 12 week (week 0 and week 12)
  Hemoglobin A1c (HbA1c) concentration in the blood will be measured
Change in C-reactive protein concentration | Every 12 week (week 0 and week 12)
  C-reactive protein concentration in the blood will be measured
Change in IL-6 concentration | Every 12 week (week 0 and week 12)
  IL-6 concentration in the blood will be measured
Change in TNF-alpha concentration | Every 12 week (week 0 and week 12)
  TNF-alpha concentration in the blood will be measured
Change in gut microbiome composition | Every 12 week (week 0 and week 12)
  Gut microbiome composition in the fecal will be measured
Change in short chain fatty acids concentration | Every 12 week (week 0 and week 12)
  Short chain fatty acids concentration in the fecal will be measured
Change in bile acid concentration | Every 12 week (week 0 and week 12)
  Bile acid concentration in the fecal will be measured

SECONDARY OUTCOMES:
Change in zonulin concentration | Every 12 week (week 0 and week 12)
  Zonulin concentration in the fecal will be measured
Change in calprotectin levels | Every 12 week (week 0 and week 12)
  Calprotectin concentration in the fecal will be measured
Change in appetite assessed by visual analogue scale | Every 4 week (week 0, week 4, week 8 and week 12)
  Visual analogue scale will be used to assess appetite.
Change in sleep quality by questionnaire | Every 4 week (week 0, week 4, week 8 and week 12)
  Questionnaire will be used to assess sleep quality
Change in weight and height | Every 4 week (week 0, week 4, week 8 and week 12)
  Weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2
Change in blood pressure | Every 4 week (week 0, week 4, week 8 and week 12)
  Systolic and diastolic blood pressure (in mmHg) will be measured by a blood pressure monitor.
Change in skin advanced glycation end products status | Every 4 week (week 0, week 4, week 8 and week 12)
  Skin advanced glycation end products status will be measured by a monitor.
Change in dietary | Every 4 week (week 0, week 4, week 8 and week 12)
  Questionnaire will be used to record dietary

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Principal Investigator — Food Science and technology, Faculty of Science, National University of Singapore
Locations (1):
- NUS Department of Food Science & Technology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on a secure website with access limited to Dr. Kim and Dr. Kim's research staff. All data will be de-identified prior to statistical analyses.